CLINICAL TRIAL: NCT03737175
Title: Endarterectomy vs Stenting in Chinese Asymptomatic Carotid Stenosis Patients: Prospective, Multiple Center, Randomized Controlled Trail
Brief Title: Endarterectomy vs Stenting in Chinese Asymptomatic Carotid Stenosis Patients
Acronym: ESCALATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Changzheng Hospital (Other); China-Japan Friendship Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Yong-Quan Gu, Prof., Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: china carotid
Record Dates: First submitted 2018-11-06; First posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Carotid Stenosis
MeSH Terms: conditions — Carotid Stenosis | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carotid Artery Stenting group (Experimental): Carotid Artery Stenting
  Interventions: Procedure: Carotid Artery Stenting
- Carotid Endarterectomy group (Active Comparator): Carotid Endarterectomy
  Interventions: Procedure: Carotid Endarterectomy

INTERVENTIONS:
Procedure: Carotid Artery Stenting — Carotid Artery Stenting
  Arms: Carotid Artery Stenting group
Procedure: Carotid Endarterectomy — Carotid Endarterectomy
  Arms: Carotid Endarterectomy group

SUMMARY:
Endarterectomy vs Stenting Asymptomatic Carotid stenosis patients to verify the efficacy and safety.

DETAILED DESCRIPTION:
Endarterectomy vs Stenting Asymptomatic Carotid stenosis patients to verify the efficacy and safety.Study Design is a prospective, multiple center, randomized controlled trail.600 cases enrollment predict，each group including carotid artery stenting and carotid endarterectomy 300 cases.Follow-up period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

Clinical Criteria

1. Age≥50 years，sex unlimited；
2. Asymptomatic carotid stenosis ，ie no transient ischemic attack、stroke or other related neurological symptom caused by carotid stenosis in the past 6 months.(Only the clinical manifestations of dizziness or mild headache are considered asymptomatic carotid stenosis.)；
3. The patient understands the trial objective，understands and accepts the duration of the study，is able and willing to comply with all requirements，including follow-up and evaluation of it, voluntarily participates in the study and signs Informed Consent Form.

   Anatomy Criteria
4. Internal carotid artery independent disease.（ Involving or not involving adjacent common carotid arteries is permitted.）；
5. Carotid stenosis satisfies one of the following criteria ：

   1. Ultrasonography suggests stenosis ≥ 70%，or angiography showed stenosis ≥ 60%；
   2. Ultrasonography suggests stenosis < 70%，but angiography or other examination showed stenosis in an unstable state；
6. Patients with bilateral carotid stenosis, the treatment time for target vessel contralateral vessels is required 30 days before enrollment or 30 days after completion of study procedure；
7. The stent can reach the site of lesion smoothly as expected.

Exclusion Criteria:

* Clinical Criteria

  1. Patients with progressive stroke in the past 3 months or recent (Within 7 days)， CT or MRI suggested that the lesion is large，and may be with the risk of hemorrhagic transformation；
  2. Patients with anesthesia contraindications；
  3. Serious ipsilateral stroke occurred in the past and may confuse the judgment of the study endpoint；
  4. Patients with severe dementia；
  5. Patients with spontaneous intracerebral hemorrhage in the past 12 months；
  6. Large size of cerebral infarction or myocardial infarction occurred within 30 days ；
  7. Patients with large intracranial aneurysms (diameter> 5mm)，and cannot be treated in advance or contemporaneous；
  8. Chronic total occlusion without obvious cerebral ischemia symptoms；
  9. Hemoglobin <100 g/l， Platelet count <125×109/L， INR>1.5， Bleeding time > 1 min，patients with exceeding the upper limits of normal，or heparin-related thrombocytopenia；
  10. Patients unable to perform normal angiographic evaluation or unsafe percutaneous puncture point；
  11. Patients with neurologic disorder that caused transient or permanent neurological deficits within 2 years before the surgery and can not be identified with transient ischemic attack or stroke；
  12. Patients with other cardiac emboli sources, such as left ventricular aneurysm, intraluminal filling defect, cardiomyopathy, aortic or mitral prosthetic heart valve, calcific aortic stenosis, infective endocarditis, mitral stenosis, atrial septal defect, atrial septal aneurysm, or left atrial myxoma；
  13. Recent gastrointestinal bleeding and affects antiplatelet therapy；
  14. Surgical contraindications or patients with high risk of surgery defined as having any of the following： It is known that two or more proximal or main coronary artery stenosis ≥70%, untreated or unable to pass； Ejection fraction <30% or New York Heart Association (NYHA) functional class III or higher； Unstable angina，ie angina at resting state and electrocardiogram changes； Currently waiting main organ transplants (ie heart, lung, liver, kidney), or are doing relevant evaluate； Malignant tumor or respiratory insufficiency, life expectancy < 5 years or forced expiratory volume at one second < 30% (predicted)； Dialysis-dependent renal failure； Poor control of diabetes, fasting blood glucose >22mmol/L and ketone body > +2； Need to perform other general anesthesia during the same period；
  15. There may be one or more anatomical conditions affecting the normal operative approach in patients with contraindications for carotid endarterectomy operation； there may be one or more anatomic situations to increase the risk of adverse events in patients with high operative risk；including： Neck radiation therapy history； Radical neck surgery history； Inoperable lesions (ie more than C2 lesions)； Spinal brake - unable to bend neck, or kyphotic deformity； Symptomatic dissection of the carotid siphon below； Common carotid artery opening lesion；present tracheotomy； Contralateral recurrent laryngeal nerve paralysis； Previously performed ipsilateral carotid endarterectomy，intracranial or subclavian arterial bypass surgery； Contralateral carotid artery occlusion； Lesions series； Severe long segment calcification of the carotid artery； Inaccessible lesions by endoluminal methods (Severe distortion of the aortic arch branch, no suitable introduction of arteries, aortic arch anatomy special）；
  16. Investigators consider the patient inappropriate to participate in this clinical trial；
  17. Those who participated in clinical trials of other drugs or medical devices before the inclusion did not reach the end of the time limit.

      Angiography criteria
  18. Severe vascular tortuosity, or anatomical conditions may affect the safe locomotion of guide catheter, guide sheath or stent；
  19. Patients with ipsilateral carotid artery stenting or having a graft；
  20. Patients with severe or extensive arteriosclerosis, involving the aortic arch and the proximal common carotid artery, causing locomotion danger of guide catheter or guide sheath；
  21. Carotid endarterectomy contraindications by angiography：severity of intracranial or extracranial arterial stenosis that exceeds target lesions; cerebrovascular arteriovenous malformations; or other contraindications;
  22. Patients with contralateral carotid artery stenosis, are expected to be performed within 30 days of the perioperative period of the study；
  23. Occlusion.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of composite endpoints of myocardial infarction, stroke, and any death | 30 days
  Incidence of composite endpoints of myocardial infarction, stroke, and any death at 30 days follow up

SECONDARY OUTCOMES:
Surgery success rate | 1 day
  Surgery success rate
Rate of complications | 30 days
  Rate of complications within 30 days, complications include：Cranial nerve and peripheral nerve injury, vascular injury, non cerebral hemorrhage, wound complications as neck incision or related to puncture site, and other (such as anesthesia) complications；
Incidence of myocardial infarction | 30 days
  Incidence of myocardial infarction at 30 days follow up;
Incidence of Ipsilateral stroke | 30 days
  Incidence of Ipsilateral stroke at 30 days follow up;
Incidence of Bilateral stroke | 30 days
  Incidence of Bilateral stroke at 30 days follow up；
Incidence of ipsilateral stroke | 12 months
  Incidence of ipsilateral stroke at 12 months follow up；
Carotid restenosis rate | 12、24 months
  Carotid restenosis rate at 12、24 months follow up；
Incidence of target lesion revascularization | 6、12、24 months
  Incidence of target lesion revascularization at 6、12、24 months follow up；
Incidence of composite endpoints of myocardial infarction, stroke, and any death | 6、12、24 months
  Incidence of composite endpoints of myocardial infarction, stroke, and any death at 6、12、24 months follow up；
Incidence of major stroke and minor stroke | 6、12、24 months
  Incidence of major stroke and minor stroke at 6、12、24 months follow up；
Surgical time | Through hospital stay，an average of 10days
  Surgical time
Hospitalization days | Through hospital stay，an average of 10days
  Hospitalization days
Hospitalization fees | Through hospital stay，an average of 10days
  Hospitalization fees

CONTACTS AND LOCATIONS:
Overall Officials: YongQuan Gu YQ Gu, Prof., Principal Investigator — Xuanwu Hospital, Beijing
Locations (6):
- China (6):
  - Sino-Japanese Friendship Hospital, Beijing
  - Shanghai Changhai Hospital, Shanghai
  - Shanghai ChangZheng Hospital, Shanghai
  - Zhongshan Hospital affiliated to Fudan University, Shanghai
  - The first affiliated Hospital of Xi ' an Jiaotong University, Xi'an
  - The first affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Giles MF, Rothwell PM. Risk of stroke early after transient ischaemic attack: a systematic review and meta-analysis. Lancet Neurol. 2007 Dec;6(12):1063-72. doi: 10.1016/S1474-4422(07)70274-0. Epub 2007 Nov 13. PMID 17993293
- [Background] North American Symptomatic Carotid Endarterectomy Trial Collaborators; Barnett HJM, Taylor DW, Haynes RB, Sackett DL, Peerless SJ, Ferguson GG, Fox AJ, Rankin RN, Hachinski VC, Wiebers DO, Eliasziw M. Beneficial effect of carotid endarterectomy in symptomatic patients with high-grade carotid stenosis. N Engl J Med. 1991 Aug 15;325(7):445-53. doi: 10.1056/NEJM199108153250701. PMID 1852179
- [Background] MRC European Carotid Surgery Trial: interim results for symptomatic patients with severe (70-99%) or with mild (0-29%) carotid stenosis. European Carotid Surgery Trialists' Collaborative Group. Lancet. 1991 May 25;337(8752):1235-43. PMID 1674060